CLINICAL TRIAL: NCT06368167
Title: A Phase II, Single-arm, Open-label, Multicenter Study on the Efficacy of SHR2554 in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: A Phase II Study of SHR2554 in Patients With Relapsed or Refractory Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-202
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR2554 (Experimental)
  Interventions: Drug: SHR2554

INTERVENTIONS:
Drug: SHR2554 — SHR2554

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR2554 in Patients with Relapsed or Refractory Follicular Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥18 years
2. Histologically confirmed follicular lymphoma
3. Eastern Cooperative Oncology Group performance status (ECOG PS) score ≤2
4. Life expectancy ≥ 12 weeks
5. Treated with CD20 antibody, refractory to or relapse from prior anti-cancer therapies
6. Have measurable lesions
7. The subject is willing and able to comply with the visit schedule, dosing schedule, laboratory tests, and other clinical study procedures

Exclusion Criteria:

1. Have been treated with a compound of the same machanism;
2. Accompanied by central nervous system infiltration;
3. Received autologous stem cell transplantation within 60 days before signing the agreement, and received allogeneic stem cell transplantation or CAR-T therapy within 90 days;
4. Underwent major surgery or experienced severe trauma within 4 weeks prior to the first dose of the investigational drug
5. Known active infection
6. History of clinically severe cardiovascular diseases
7. Have other malignancies within 5 years prior to screening Pregnant or lactating women
8. The subject is unable to swallow, or has a history of active gastrointestinal inflammation, chronic diarrhea, known diverticulosis, or a history of gastrectomy or gastric banding that affects drug absorption.
9. The subject is taking a known medium or strong CYP inducer.
10. Based on the investigator's judgment, there are objective conditions that may prevent the subject from completing the study as planned or the subject has other factors, concomitant diseases, concomitant treatments, or abnormal laboratory findings that may lead to early study termination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by independent review committee (IRC) | around 1 year
  percentage of patients who achieve completes response(CR) or partial response(PR) in the study

SECONDARY OUTCOMES:
ORR assessed by investigator | around 1 year
  percentage of patients who achieve CR or PR in the study
Progression free survival | around 1 year
  time from the first dose of SHR2554 to the first disease progression(PD) or death
Time to Response | around 4 months
  time from the first dose of SHR2554 to first CR or PR
Duration of response | around 1 year
  time from the first CR or PR to the first PD or death
Overall survival | around 5 years
  time from the fist dose of SHR2554 to death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China